CLINICAL TRIAL: NCT07380555
Title: A Multicenter, Cluster-randomized, Controlled Study Evaluating the Effectiveness and Safety of Artificial Intelligence(AI)-Assisted Medical Treatment Decision Support System Compared to Conventional Care in HFrEF Patients
Brief Title: The Effectiveness and Safety of Artificial Intelligence(AI)-Assisted Medical Treatment Decision Support System Compared to Conventional Care in HFrEF Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2025-392R2
Record Dates: First submitted 2026-01-12; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HF-rEF)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Guided Group (Experimental): patients in this group will receive medication recommendations from an AI system based on patient health data.
  Interventions: Device: artificial intelligence (AI) decision support system
- Standard Care Group (No Intervention): patients in this group will receive medications as normally plan, without AI assistance.

INTERVENTIONS:
Device: artificial intelligence (AI) decision support system — According to the data uploaded by patients, drug treatment plan were generated based on a prespecified AI-assisted decision-making system, which were reviewed by researchers and sent to patients
  Arms: AI-Guided Group

SUMMARY:
This clinical trial aims to find out if using an artificial intelligence (AI) decision support system can help doctors better manage medications for people with heart failure with reduced ejection fraction (HFrEF). The main goal is to see if this approach can lower the chance of patients being hospitalized for heart failure or dying from heart-related causes compared to standard care.

About 1,200 participants from 60 hospitals will take part in this study. The hospitals, not the individual patients, are randomly assigned to one of two groups:

AI-Guided Group: Doctors at these hospitals will receive medication recommendations from an AI system based on patient health data.

Standard Care Group: Doctors at these hospitals will manage medications as they normally would, without AI assistance.

All participants will have regular check-ups, both remotely every 30 days and in-person at 3, 6, and 12 months. The study will last about 12 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Patients diagnosed with HF in hospital and discharged on medical orders;
3. LVEF≤40% detected by echocardiography within 1 month before enrollment;
4. Signed informed consent is obtained.

Exclusion Criteria:

1. Patients who are unable or unsuitable for follow-up.
2. Patients with poor compliance, presenting a risk of switching study groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite endpoint of heart failure rehospitalization or cardiovascular death | 12 months
  The occurrence of the first event of either hospitalization due to worsening heart failure or death from a cardiovascular cause.

SECONDARY OUTCOMES:
All-cause rehospitalization | From enrollment to 12 months follow-up
  Hospitalization for any cause
Change from baseline in Left Ventricular End-Diastolic Diameter (LVEDD) | Baseline and 12 months
  The absolute change in the internal diameter of the left ventricle at the end of its filling phase (millimeters, mm).
Cardiovascular mortality | From enrollment to 12 months follow-up
  Death due to cardiovascular causes
All-cause mortality | From enrollment to 12 months follow-up
  Death from any cause
From enrollment to 12 months follow-up | From enrollment to 12 months follow-up
  The total count of heart failure-related hospitalizations per participant.
Change from baseline in NT-proBNP level | Baseline and 12 months
  The absolute or relative change in the N-terminal pro-brain natriuretic peptide level from the start of the study to the follow-up time point.
Change from baseline in Left Ventricular Ejection Fraction (LVEF) | Baseline and 12 months
  The absolute change in the percentage of blood pumped out of the left ventricle with each contraction.
Change from baseline in Left Ventricular End-Diastolic Diameter (LVEDD) | Baseline and 12 months
  The absolute change in the internal diameter of the left ventricle at the end of its filling phase(millimeters, mm).
Change from baseline in quality of life score as assessed by the EQ-5D | Baseline and 12 months
  The change in the score from the EQ-5D quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data collected in this study are not currently planned for sharing due to privacy and ethical constraints. However, reasonable requests for de-identified data will be considered by the corresponding investigator upon submission of a methodologically sound proposal.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT07380555/Prot_SAP_000.pdf